CLINICAL TRIAL: NCT00143858
Title: Assessment of the Clinical Utility of Non Invasive Peripheral Signal Averaged Pulse Volume
Status: Completed | Type: Observational
Sponsor: University of Medicine and Dentistry of New Jersey (Other)
Responsible Party: Sebastian T. Palmeri, MD -- Principal Investigator, UMDNJ-Robert Wood Johnson Medical School
Organization: Rutgers, The State University of New Jersey (Other)
Other Study IDs: 4301; investigator initiated
Record Dates: First submitted 2005-08-31; First posted 2005-09-02 (Estimated); Last update posted 2009-08-11 (Estimated); Status verified 2009-08

CONDITIONS: Peripheral Vascular Response
Keywords: Peripheral Pulse Volume

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Pulse Volume Measurement — patients will wear a newly designed calf monitor that will be hooked up to a computer that will monitor leg peripheral pulse volumes which will then be correlated to pressures obtained with Swan Ganz monitoring. The calf monitor is gut two bands with sensors that are wrapped around the ankle and below the knww

SUMMARY:
The purpose of this study is to determine the clinical usefulness of measuring the heart's pumping ability by measuring the Peripheral Pulse Volume (PPV).

DETAILED DESCRIPTION:
Peripheral Pulse Volume (PPV) is the change in the volume of a limb that occurs when blood passes through the limb. The limb also acts as an electrical conductor whose electrical impedence changes with limb geometry and volume. Each time the heart beats, the volume of the limb segment changes, and therefore its electrical impedence changes. A plethysmograph can be used to measure volume changes of a part of the body by producing a plethysmographic waveform. Selectively capturing a number of these plethysmographic wave forms with acceptable noise levels and averaging them using the EKG as a reference-timing signal generate a highly reproducible pulse volume signal. Signal averaged pulse volume measurement will be obtained non-invasively from the lower extremities of patient volunteers. A disposal non-occluding electrical monitoring strap will be applied to the calf of each patient. Changes in the calf's size/volume caused by changes in the patient's cardiac output and calf blood flow will result in electrical impedance changes. These changes will be recorded by an analog admittance plethysmograph attached to the lower extremity strap. The analog plethysmograph is coupled to a digital computer for signal enhancement and measurement.

ELIGIBILITY:
Inclusion Criteria

* Coronary care unit patients with indwelling right heart (Swan Ganz) catheters with or without intraaortic balloon assist pumping devices.
* Congestive Heart Failure patients on and off various therapeutic inotropic agents with or without indwelling heart catheters
* Cardiac catheterization laboratory patients undergoing prophylactic IABP in the presence of left main or diffuse unstable CAD
* Chronic renal failure patients undergoing hemodialysis.
* Peripheral Vascular Disease patients
* Patients undergoing Tilt Table Testing
* Any patients undergoing right heart catheterization Exclusion criteria -- Non specified

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient who are having a right heart catherization done for other diagnostic purposes or patient in the critical care units who have Swan Ganz catheters in place for other medical management
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2004-09; Study Completion 2007-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sebastian Palmeri, MD, Principal Investigator — Rutgers, The State University of New Jersey
Locations (1):
- Robert Wood Johnson University Hospital, New Brunswick, New Jersey, United States

REFERENCES:
- [Background] Marks LA. Digital enhancement of the peripheral admittance plethysmogram. IEEE Trans Biomed Eng. 1987 Mar;34(3):192-8. doi: 10.1109/tbme.1987.325944. No abstract available. PMID 3570309